CLINICAL TRIAL: NCT05069285
Title: A Randomized Controlled Trial Comparing a Self-help Book Focusing on Cognitive Behavioral Therapy for Insomnia With Standard Sleep Hygiene Advice Among Patients Using Hypnotics
Brief Title: A Self-help Book for Insomnia Compared With Sleep Hygiene Advice in Patients Using Sleep Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Bjorn Bjorvatn, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PraksisNettRCT2022
Record Dates: First submitted 2021-09-23; First posted 2021-10-06 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Hypnotic; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-help book (Experimental): A self-help book for insomnia (written in Norwegian)
  Interventions: Other: self-help book
- Sleep hygiene advice (Active Comparator): A sheet of paper with standard sleep hygiene advice
  Interventions: Other: sleep hygiene advice

INTERVENTIONS:
Other: self-help book — information and advice given in the self-help book
  Arms: Self-help book
Other: sleep hygiene advice — information and advice given on the sheet of paper with sleep hygiene
  Arms: Sleep hygiene advice

SUMMARY:
The aim is to assess whether a self-help book for insomnia will improve sleep and reduce hypnotic use among patients on sleep medications.

DETAILED DESCRIPTION:
This study is a randomized controlled trial evaluating the effect of a self-help book for insomnia compared to the effect of sleep hygiene advice in patients using sleep medications. 150 patients will be randomized to receive either the book (75 patients) or the sleep hygiene advice (75 patients). Patients will fill questionnaires about sleep and health problems at baseline and after 3-6 months after receiving the written material. The main aims are to assess whether a self-help book is more effective in reducing sleep medication use and sleep problems.

ELIGIBILITY:
Inclusion Criteria:

- Use of sleep medications on prescription or OTC during the last 6 months

Exclusion Criteria:

- Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Use of hypnotics assessed as days per week | 3-6 months
  Self-reported sleep medication use (days of use per week,0-7)
Insomnia severity assessed with Insomnia Severity Index | 3-6 months
  Self-reported sleep problems on the validated Insomnia Severity Index (0-28), with higher scores indicating worse sleep
Insomnia severity assessed with Bergen Insomnia Scale | 3-6 months
  Self-reported sleep problems on the validated Bergen Insomnia Scale (0-42), with higher scores indicating worse sleep

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Bjorvatn, MD PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No